CLINICAL TRIAL: NCT06803407
Title: Investigation of the Effectiveness of a Home Exercise Program in Individuals With Temporomandibular Joint Disc Displacement With Reduction
Brief Title: Investigation of the Effectiveness of a Home Exercise Program
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nurhayat KORKMAZ, Research assistant, Karadeniz Technical University
Other Study IDs: KTU-FTR-2024/7
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Joint Disc Displacement
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1 study group: Home exercise group and patient education
  Interventions: Other: Home exercise; Other: Patient education
- Group 2 control group: Only patient education
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Home exercise — The study group will be given exercises that include temporomandibular joint and neck as a home exercise program.
  Groups: Group 1 study group
Other: Patient education — Information about the disease and symptoms, chewing recommendations, dietary changes, parafunctional habits, activities to avoid, posture training

SUMMARY:
The purpose of this study is to examine the effects of a home exercise program on individuals with temporomandibular joint disc displacement with reduction. Participants will be assessed at baseline and again after a four-week home exercise program.

DETAILED DESCRIPTION:
Participants who meet the inclusion criteria will be randomly divided into 2 groups. The first group, called the study group, will receive a home exercise program and patient education. The second group, called the control group, will receive only patient education. Participants will be assessed at baseline and again after a four-week home exercise program.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 65 years,
* who have had complaints related to TMJ for at least 3 months,
* who have been diagnosed with Temporomandibular joint disc displacement with reduction as a result of clinical and radiological evaluation by a dentist

Exclusion Criteria:

* Those with cognitive problems,
* any systemic joint or muscle disease (e.g. fibromyalgia, rheumatoid arthritis),
* serious systemic diseases,
* any neurological disorder (e.g. trigeminal neuralgia),
* pregnancy, breastfeeding,
* who have previously been treated for TMJ or orofacial muscle pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Temporomandibular joint disc displacement with reduction
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Range of motion | an average one month
  Range of motion of temporomandibular joint

SECONDARY OUTCOMES:
Numeric Pain scale | an average one month
  Pain severity assessment
Mandibular Function Impairment Questionnaire | an average one month
  Assessment of mandibular function

CONTACTS AND LOCATIONS:
Overall Officials: Nurhayat korkmaz, Msc, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No